CLINICAL TRIAL: NCT01313247
Title: Optimizing Medication for Cancer Pain. The Effect of Paracetamol. A Clinical and Pharmacological Trial to Research Whether Paracetamol Gives an Additional Effect on Pain Relief When the Patient is Treated With High Doses of Opioids
Brief Title: Paracetamol for Cancer Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haraldsplass Deaconess Hospital (Other)
Responsible Party: Jan Henrik Rosland, professor, Haraldsplass Deaconess Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Par 06-0045
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Advanced Cancer; Opioid Use, Unspecified
Keywords: Paracetamol; opioids; cancer pain
MeSH Terms: conditions — Cancer Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo pills (Placebo Comparator): Placebo tablets resembling paracetamol 500 mg are given as alternative 2 tablets 4 times daily
  Interventions: Drug: placebo tablets
- oral paracetamol 4 g daily (Active Comparator): Patients are given 2 tablets of 500 mg paracetamol on a regular basis 4 times daily
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: paracetamol — 1000 mg 4 times daily
  Other Names: Acetaminophen
  Arms: oral paracetamol 4 g daily
Drug: placebo tablets — Placebo pills eqv paracetamol are given 2 tablets 4 times daily instead of paracetamol
  Other Names: Suger pills
  Arms: Placebo pills

SUMMARY:
Randomised, double-blind placebo controlled cross-over trial

Main goal:

Optimize the medical pain treatment for patients with advanced cancer disease

Study goal:

Measure paracetamol's additional analgesic effect in a situation where the patient is concomitantly treated with oral opioids eqv. morphine > 100 mg/d.

DETAILED DESCRIPTION:
National multicenter study with an intention to include 50 patients. 6 days treatment, 3d in each arm. Mean pain score last 24 h: NRS =/> 4 All drug treatment constant during the study period. The participants are allowed to take as much rescue opioids as necessary to have adequate relief.

Paracetamol/ placebo given orally 1000 mg x 4 daily, three days in each arm, direct crossover.

Daily scoring of pain relief, ESAS, overall satisfaction and rescue medication.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years) of both sexes
* Diagnosed with advanced cancer disease
* Ongoing medicinal pain relief treatment in stable dosing with oral opiates equivalent to > 100 mg oral morphine daily
* NRS median pain score last 24 hrs > 4
* Able to take tablets (paracetamol) orally

Exclusion Criteria:

* Mental or physical deficiency precluding data collection.
* Reduced liver function judged with bilirubin, INR and transaminases
* Anticoagulation with warfarin
* Ongoing use of NSAIDs or 5-HT3 antagonists, or use of such drugs last week
* Ongoing palliative radiation treatment or radiation treatment during the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Pain reduction caused by paracetamol 4g/d | Last day in each 3 days study period
  Pain reduction in the active paracetamol arm, compared to placebo, corrected for difference in rescue medication intake.

SECONDARY OUTCOMES:
Overall satisfaction with the pain treatment | End of each 3 days study period
  Total ESAS score Sweating during nighttime general wellbeing

CONTACTS AND LOCATIONS:
Overall Officials: Jan Henrik Rosland, MD, PhD, Principal Investigator — Haraldsplass Deaconess Hospital
Locations (1):
- Haraldsplass Deaconess Hospital, Bergen, Norway